CLINICAL TRIAL: NCT06686719
Title: Comparison of Post Facilitation Stretch, Post Isometric Relaxation and Myofascial Release on Lower Limb Spasticity in Spastic Cerebral Palsy.
Brief Title: Post Facilitation Stretch, Post Isometric Relaxation and Myofascial Release in Spastic Cerebral Palsy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRAHS/REC/MS-PT/01942
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Spastic Diplegia Cerebral Palsy
Keywords: Spastic Cerebral Palsy; Myofascial; Spasticity
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic; Cerebral Palsy; Muscle Spasticity | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post Facilitation group (Experimental): subjects are asked to isometrically contract the hamstring and calf using 30 % of the strength for 15 seconds by attempting to push the leg back toward the therapist and relax. The therapist then passively stretched the muscle until a mild stretch sensation was reported. The stretch was held for another 10 seconds. This sequence will repeat 5 times on each subject in the group.
  Stretching of the hip flexors, adductors and plantarflexor muscles. Functional training includes bridging, kneeling, sit to stand
  Interventions: Other: Post Facilitation
- Post Isometric Relaxation (Active Comparator): Subjects are asked to isometrically contract the hamstring and calf using 25 % of the strength for 7-10 seconds by attempting to push the leg back toward the therapist and relax. After relaxation, the therapist further extends the knee for 3 to 5 seconds. This sequence will repeat 5 times on each subject in the group.
  Stretching of the hip flexors, adductors and plantarflexor muscles. Functional training includes bridging, kneeling, sit to stand.
  Interventions: Other: Post Isometric Relaxation
- Myofascial Release (Active Comparator): MFR for Hamstring muscle will be given with patient in prone position with 120 second hold. For giving the MFR, the thumb of the therapist will be allowed to sink in to the central portion of the hamstring. It will held for 120 seconds to allow the tissue to soften and then myofascial structures will spread in a lateral direction until feeling of first fascial barrier. MFR will be performed for 15 mins.
  Interventions: Other: Myofascial Release

INTERVENTIONS:
Other: Post Facilitation — For hamstring muscle, the patient positioned in supine with hip and knee flexed to mid- range. For calf muscle, the patient positioned in supine with straight leg. Now therapist ask the subjects to isometrically contract the hamstring and calf using 30 % of the strength for 15 seconds by attempting to push the leg back toward the therapist and relax. The therapist then passively stretched the muscle until a mild stretch sensation was reported. The stretch was held for another 10 seconds. This sequence will repeat 5 times on each subject in the group.
  Stretching of the hip flexors, adductors and plantar flexors. Functional training includes bridging, kneeling and sit to stand.
  Arms: Post Facilitation group
Other: Post Isometric Relaxation — For hamstring muscle, the patient positioned in supine with hip and knee flexed. For calf muscle, the patient positioned in supine with straight leg. Now therapist ask the subjects to isometrically contract the hamstring and calf using 25 % of the strength for 7-10 seconds by attempting to push the leg back toward the therapist and relax.After relaxation, the therapist further extends the knee for 3 to 5 seconds.. This sequence will repeat 5 times on each subject in the group.
  Stretching of the hip flexors, adductors and plantar flexors. Functional training includes bridging, kneeling and sit to stand.
  Arms: Post Isometric Relaxation
Other: Myofascial Release — MFR for Hamstring muscle will be given with patient in prone position with 120 second hold. For giving the MFR, the thumb of the therapist will be allowed to sink in to the central portion of the hamstring. It will held for 120 seconds to allow the tissue to soften and then myofascial structures will spread in a lateral direction until feeling of first fascial barrier. MFR will be performed for 15 mins.
  Stretching of the hip adductors, hip flexors and plantar flexors. Functional training includes kneeling, bridging and sit to stand.
  Arms: Myofascial Release

SUMMARY:
The purpose of the study is to compare the effect of Post Facilitation Stretch, Post Isometric Relaxation and Myofascial Release on Lower Limb Spasticity in Spastic Cerebral Palsy. A randomized control trial was conducted at PAF School for PSN NUR KHAN Rawalpindi. The sample size was 30 calculated through G-Power tool. The participants were divided into three interventional groups each having 10 participants. The study duration was six months. Sampling technique applied was Convenient sampling for recruitment and group randomization using lottery method. Only 8 to 18 years Spastic Dipelgic CP children with Modified Asworth Scale having score 1, 1+ and 2 were included in the study. Tools used in this study are Goniometer, Modified Ashworth Scale, Active knee extension test, Weight bearing lunge test. Data was collected before and immediately after the application of interventions. Data analyzed through SPSS version 26.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a disorder affecting movement, resulting from permanent damage to posture and motor development during fetal or infant brain development, caused by non-progressive disturbances. CP affecting about 1 in 500 children with an estimated prevalence of 17 million people worldwide. In CP, spasticity is often regarded to be the most common motor impairment. Spastic cerebral palsy stands out as the predominant subtype, constituting 77% of all cases, with bilateral spastic cerebral palsy dominating the spastic group (70%). Spasticity is only one of several components of the upper motor neuron (UMN) syndrome. Spasticity is a form of hypertonia due to hyperexcitable tonic stretch reflexes. Adult CP reported that 77% of CP children were having problems with spasticity. Hypertonicity resulting in abnormal movement patterns in both gross motor function and manual abilities in the children with CP.

Traditionally the treatment of tightness in children with spasticity has consisted primarily of techniques which involve static stretching, strengthening of the antagonistic muscles, use of orthosis and postural education etc. Some authorities also recommend Myofascial release to cause elongation of the spastic muscle with a component of tightness. Myofascial therapy can be defined as "the facilitation of mechanical, neural and psycho physiological adaptive potential as interfaced by the myofascial system". Akta Bhalara et al (2014) concluded in a study that myofascial release is effective in reducing spasticity in children suffering from spastic diplegic cerebral palsy. A study conducted in 2018 proved that myofascial release is effective in reducing spasticity of hamstring muscle and improves range of motion in spastic diplegic cerebral palsy. Ujwal Bhattacharya et al (2017) in a study concluded that MFR and passive stretching is effective in reducing spasticity and improving range of motion in spastic diplegic Cerebral Palsy.

Fred Mitchell first described MET in 1948 as a type of osteopathic manipulative diagnosis and treatment, primarily utilized to address somatic dysfunction, particularly issues such as reduced range of motion, muscular hypertonicity, and pain. MET involves the use of two physiological phenomena: Post Isometric Relaxation and Reciprocal Inhibition. Post Isometric Relaxation is a technique that was later developed by Karel Lewitt . Post Isometric Relaxation (PIR) is the effect of the decrease in muscle tone in a single or group of muscles, after a brief period of submaximal isometric contraction of the same muscle.

Preeti Gazbare et al ( 2018) conducted a Comparative Study On The Effect of Myofascial Release Over Post Isometric Relaxation On Calf Muscle Tone in Spastic Diplegic Cerebral Palsy and concluded that both MFR and PIR are equally effected in reducing calf muscle tone in spastic Cerebral Palsy. PIR improves better flexibility and decrease tightness of hamstring muscle as compared to static stretching. MET improves the independent mobility of stroke patients with hemiplegia enhances balance and stability. Janstephan T (2015) conducted a study to evaluate the effectiveness of neurodevelopment therapy with post isometric relaxation for lower extremity to improve functional ability in children with spastic diplegic cerebral palsy. The result suggested that neurodevelopmental therapy along with muscle energy technique improved the functional ability in children with spastic diplegic cerebral palsy.

Post Facilitation Stretch (PFS) is a technique developed by Janda.This technique is more aggressive than PIR but is also based on the concept of autogenic inhibition. Post facilitation stretching is a MET technique which uses postisometric relaxation. The term refers to the effect of the subsequent relaxation experienced by a muscle after an isometric contraction has been performed. The effect of a sustained contraction on the Golgi tendon organs seems pivotal, since their response to such a contraction seems to be set the tendon and the muscle to a new length by inhibiting it. A study concluded that Post Facilitation Stretching is effective in increasing Flexibility of tight hamstring muscles. A study concluded that post facilitation stretch is effective in reducing pain and improving muscle length. A study in published in 2024 compared the effect of the muscle energy technique (MET) and stretching technique on ankle dorsiflexion passive range of motion, balance, and gait ability of stroke patients with limited ankle dorsiflexion. And concluded that MET and Stretching both are effective in improving range of motion , balance and gait ability of stroke patients with limited ankle dorsiflexion.

The rationale for this study is that Post-facilitation stretch relaxation (PFSR) is proposed as an effective intervention for reducing lower limb spasticity in spastic cerebral palsy. By combining passive stretching with relaxation techniques post- facilitation, PFSR aims to decrease muscle tone and improve range of motion. This approach is individualized, often integrated with other therapies, and emphasizes patient education for long term management.

ELIGIBILITY:
Inclusion Criteria:

* Spasticity score of less than 3 on MAS
* Known cases of Spastic diplegic cerebral palsy.
* Children who follow commands.

Exclusion Criteria:

* Epilepsy history
* hip or spinal deformities
* Severe contractures, joint dislocations
* Discrepancy in leg length
* Recent orthopedic surgery
* Children with cognitive impairment.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-12-03 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Four Weeks
  Changes from the baseline spasticity measured with help of modified ashworth scale
Range of motion | Four Weeks
  Changes from baseline range of motion of hip, knee and ankle will be measured with help of goniometer.

SECONDARY OUTCOMES:
Active Knee Extension Test | Four Weeks
  Changes from the baseline hamstring tightness will be measured with active knee extension test
Weight Bearing Lunge Test | Four Weeks
  Changes from the baseline calf tightness will be measured with weight bearing lunge test

CONTACTS AND LOCATIONS:
Overall Officials: Ammanullah Nazir, PHD*, Principal Investigator — Riphah International University Islamabad
Locations (1):
- PAF School For PSN NUR KHAN, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No